CLINICAL TRIAL: NCT01181700
Title: An Open Study To Estimate The Plasma Pharmacokinetics Of PF-00241939 Administered Via Oral Inhalation Using Dry Powder Inhalers
Brief Title: A Study To Estimate The Time Course Of PF-00241939 Concentration In The Blood After Dosing With Oral Inhalation From Dry Powder Inhalers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: B0871015
Record Dates: First submitted 2010-08-11; First posted 2010-08-13 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Pharmacokinetics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Treatment A (Experimental)
  Interventions: Drug: Treatment A
- Treatment B (Experimental)
  Interventions: Drug: Treatment B
- Treatment C (Experimental)
  Interventions: Drug: Treatment C
- Treatment D (Active Comparator)
  Interventions: Drug: Treatment D
- Treatment E (Active Comparator)
  Interventions: Drug: Treatment E
- Treatment F (Active Comparator)
  Interventions: Drug: Treatment F
- Treatment G (Active Comparator)
  Interventions: Drug: Treatment G

INTERVENTIONS:
Drug: Treatment A — PF-00241939 300 ug using inhaler A
  Arms: Treatment A
Drug: Treatment B — PF-00241939 300 ug using inhaler A
  Arms: Treatment B
Drug: Treatment C — PF-00241939 300 ug using inhaler A
  Arms: Treatment C
Drug: Treatment D — PF-00241939 300 ug using inhaler B
  Arms: Treatment D
Drug: Treatment E — PF-00241939 300 ug using inhaler B
  Arms: Treatment E
Drug: Treatment F — PF-00241939 300 ug using inhaler B
  Arms: Treatment F
Drug: Treatment G — PF-00241939 300 ug using inhaler B
  Arms: Treatment G

SUMMARY:
The purpose of this study is to investigate the time course of PF-00241939 concentrations in the blood following dosing by oral inhalation using dry powder inhalers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 21 and 55 years.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Pregnant or nursing females.
* A positive urine drug screen.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2010-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Plasma pharmacokinetic parameters: AUClast and Cmax. | 36 hours

SECONDARY OUTCOMES:
Plasma pharmacokinetic parameters: AUC24, AUCinf, Tmax and half-life. | 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0871015&StudyName=A%20Study%20To%20Estimate%20The%20Time%20Course%20Of%20PF-00241939%20Concentration%20In%20The%20Blood%20After%20Dosing%20With%20Oral%20Inhalation%20From%20Dry%20Powder%20Inha